CLINICAL TRIAL: NCT04016454
Title: Impact of Handover of Anesthesia Care on Adverse Postoperative Outcomes
Acronym: HandiCAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: Else Kröner Fresenius Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 04-AnIt-18
Record Dates: First submitted 2019-06-27; First posted 2019-07-11 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Anesthesia; Adverse Effect of Handovers of Anesthesia Care
Keywords: handover; intraoperative; anesthesia; adverse outcomes
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: In order to investigate the impact of handover of anesthesia care on adverse postoperative outcomes, patients will be assigned to the two randomization groups:
  1. Intervention group: handover of anesthesia
  2. Control group: no handover of anesthesia
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): No handover of anesthesia care
  Interventions: Procedure: Intervention
- Control group (No Intervention): Complete handover of anesthesia care

INTERVENTIONS:
Procedure: Intervention — There will be one complete handover
  Arms: Intervention group

SUMMARY:
Our goal is to conduct a prospective, national, randomized-controlled, multicenter trial to investigate the effect of handover of anesthesia care on the occurrence of adverse outcomes in the perioperative period.

DETAILED DESCRIPTION:
Intraoperative handover of anesthesia care frequently occurs in clinical routine. Communication between the two anesthesiologists plays a pivotal role for the continuation of anesthesia care. The outgoing clinician must inform the incoming clinician in a short period of time about the important pre- and intraoperative facts and about the surgery while continuing to provide patient care. Contributing factors to inadequate communication during handoffs include insufficient or misleading information, busy and distractive environment, ineffective communication methods, lack of time, lack of standardized procedures, and insufficient staffing. It is estimated that the majority of adverse events in health care involve miscommunication during the handoff between physicians and perhaps other health care practitioners (https://www.jointcommission.org/hot_topics_toc/).

The goal is to conduct a prospective, national, randomized-controlled, multicenter trial to investigate the effect of handover of anesthesia care on the occurrence of adverse outcomes in the perioperative period. The investigators hypothesizes that handover of anesthesia care does increase the risk for adverse outcomes. The primary outcome parameter is a combined endpoint consisting of all-cause mortality, readmission to any hospital, or major postoperative complications (including prolonged postoperative ventilation ≥ 48 h, major disruption of surgical wound, bleeding, pneumonia, atrial fibrillation, moderate or severe acute kidney injury, new onset of hemodialysis, cardiac arrest, myocardial infarction, sepsis, stroke, pulmonary embolism, deep venous thrombosis, shock, unplanned return to operating room) within 30 days of index surgery. Secondary endpoints are the individual criteria of the primary endpoint, hospital length of stay, ICU admission, and ICU length of stay. As the currently available data on handover of anesthesia care have not been obtained from prospective, randomized controlled trials, the results of the Handicap trial will bring new insights to anesthesia care to improve patients' outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Major surgeries with a duration of at least 2 h (requirement of postoperative admission to hospital for at least 1 night)
* ASA 3-4
* Informed consent

Exclusion Criteria:

* Previous surgery within the same surgical subgroup within the last 6 months
* Pregnancy, breastfeeding
* Patients participating in another interventional trial within the last 3 months
* Persons with any kind of dependency on the investigator or employed by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1817 (Actual)
Dates: Start 2019-06-21 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Combined endpoint consisting number of participants with all-cause mortality, readmission to any hospital or major postoperative complications | within 30 days of index surgery

SECONDARY OUTCOMES:
Number of participants with all-cause mortality | within 30 days of index surgery
Numer of participants with readmission to any hospital | within 30 days of index surgery
Number of participants with major postoperative complication | within 30 days of index surgery
  predefined postoperative complication including prolonged postoperative ventilation ≥ 48h, major disruption of surgical wound, bleeding, pneumonia, atrial fibrillation, moderate or severe acute kidney injury, new onset of hemodialysis, cardiac arrest, myocardial infarction, sepsis, stroke, pulmonary embolism, deep venous thrombosis, shock, unplanned return to operating room
Hospital length of stay | within 30 days of index surgery
Number of patients with ICU admission | within 30 days of index surgery
ICU length of stay | within 30 days of index surgery

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Meersch, MD, PHD, Principal Investigator — University Hospital Muenster, Dept. of Anesthesiology, Intensive Care and Pain Medicine
Locations (11):
- Germany (11):
  - University Hospital Aachen, Aachen
  - University Hospital Bochum, Bochum
  - Kliniken der Stadt Köln gGmbH, Klinik für Anästhesiologie und operative Intensivmedizin, Cologne
  - Klinikum Dortmund, Dortmund
  - St. Josefs-Hospital Dortmund-Hörde, Dortmund
  - Florence-Nightingale-Krankenhaus, Düsseldorf
  - Universitätsmedizin Göttingen, Klinik für Anästhesiologie, Göttingen
  - University Hospital Heidelberg, Heidelberg
  - Kliniken Maria Hilf, Mönchengladbach
  - University Hospital Muenster, Münster
  - St. Franziskus Hospital, Münster

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meersch M, Weiss R, Kullmar M, Bergmann L, Thompson A, Griep L, Kusmierz D, Buchholz A, Wolf A, Nowak H, Rahmel T, Adamzik M, Haaker JG, Goettker C, Gruendel M, Hemping-Bovenkerk A, Goebel U, Braumann J, Wisudanto I, Wenk M, Flores-Bergmann D, Bohmer A, Cleophas S, Hohn A, Houben A, Ellerkmann RK, Larmann J, Sander J, Weigand MA, Eick N, Ziemann S, Bormann E, Gerss J, Sessler DI, Wempe C, Massoth C, Zarbock A. Effect of Intraoperative Handovers of Anesthesia Care on Mortality, Readmission, or Postoperative Complications Among Adults: The HandiCAP Randomized Clinical Trial. JAMA. 2022 Jun 28;327(24):2403-2412. doi: 10.1001/jama.2022.9451. PMID 35665794